CLINICAL TRIAL: NCT04960176
Title: Development and Validation of Non-Invasive Sham Technique Using Blunted Acupuncture Needle
Brief Title: Validation of a Non-Invasive Sham Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Pınar Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 08.06.2021/31
Record Dates: First submitted 2021-07-06; First posted 2021-07-13 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Active Comparator): Acupuncture will be administered to 5 different reel acupoints. The acupoints are Du20 in head, LI4 bilateral in hands and ST36 bilateral in legs.
  Interventions: Procedure: Acupuncture
- Non-Invasive Sham Acupuncture Group (Sham Comparator): Non-invasive sham acupuncture using a blunted needle will be administered to 5 different reel acupoints. The acupoints are Du20 in head, LI4 bilateral in hands and ST36 bilateral in legs.
  Interventions: Procedure: Non-invasive Sham Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture will be applied by using 0,25x25mm needles.
  Arms: Acupuncture Group
Procedure: Non-invasive Sham Acupuncture — Non-invasive sham acupuncture will be applied by using blunted 0,25x25mm needles.
  Arms: Non-Invasive Sham Acupuncture Group

SUMMARY:
The objective of this study is to develop, describe in detail and validate a feasible, cheap and convenient non-invasive sham acupuncture technique in order to use safely and repeatedly in future studies. Additionally, the reactions of the volunteers to sham needles in different positions and in different parts of the body will be investigated.

DETAILED DESCRIPTION:
Following the Second World War, the evidence based research is the keystone of modern medicine applications. Randomized, placebo controlled and double/triple blinded clinical studies are the sine qua non of evidence based medicine. As a matter of course acupuncture which was defined as traditional and the main outcome was the clinical effects throughout the centuries, had its share form the tremendous evolution. For the past decades, studies on acupuncture are designed and prosecuted on the basis of randomized and placebo controlled trials.

In clinical trials for invasive modalities, placebo is the procedure that mimics the original procedure in order to provide objective comparison. These procedures are called as sham techniques and in acupuncture sham techniques are divided into two categories as invasive sham procedures and non-invasive sham procedures. Non-invasive sham is a technique that is designed to create a minor sensory stimulation in the absence of skin penetration using a placebo needle or any device imitating needle. In acupuncture practice it is a fact that sham procedures are non-inert and even can exert high therapeutic effect. Consequently, the main concern regarding the randomized controlled trials on acupuncture is that false negative rates might be misleadingly higher than acceptable values. The clinical therapeutic effects of non-invasive techniques are attributed to the activation of physiologic endogen systems due to the belief that acupuncture was applied although it was only sham. Non-invasive techniques need to be used in clinical trials designed to discriminate this mentioned effect from the point-specific effects of real acupuncture and non-specific effects obtained by skin penetration in invasive sham techniques.

The fact that sham techniques used in clinical studies are far from standardization inevitably increase the false negativity rates. In fact there are various techniques about non-invasive sham acupuncture. Blunted needles or plastic guide tube, nail, pencil point probe or even wooden skewers were used. Techniques are not described most of the time and majority of the studies lack standardization and validation of the non-invasive sham technique that is used. There are standard Park and Steinberger needles which were developed privately for non-invasive sham procedures. The advantage these latter needles is that the patient cannot see the application of the needle. Otherwise as in all non-invasive sham technique the needles do not penetrate the skin, the patient does not get the de chi sensation and the stimulation of the needles is not possible.

ELIGIBILITY:
Inclusion Criteria:

* The healthy attendants of patients referred to General Surgery outpatient clinic

Exclusion Criteria:

* presence of any diagnosed disease
* on any regular medication
* skin reaction on the area of planned acupuncture administration
* neurologic sequela

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Perception of Needle Penetrating the Skin | Through study completion, an average of 3 months
  Measured by a question addressing if the patient felt any penetration through the skin or not. Answer 'YES' is interpreted as sham procedure successfully mimicks real acupuncture. Answer 'NO' is interpreted as a failure of sham procedure in mimicking real acupuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Erdoğan, MD, Principal Investigator — Niğde Ömer Halisdemir University Midwifery Department
Locations (1):
- Niğde Ömer Halisdemir University Research and Training Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaptchuk TJ. Placebo Effects in Acupuncture. Med Acupunct. 2020 Dec 1;32(6):352-356. doi: 10.1089/acu.2020.1483. Epub 2020 Dec 16. PMID 33362886
- [Background] Birch S. A review and analysis of placebo treatments, placebo effects, and placebo controls in trials of medical procedures when sham is not inert. J Altern Complement Med. 2006 Apr;12(3):303-10. doi: 10.1089/acm.2006.12.303. PMID 16646730
- [Background] Lundeberg T, Lund I, Naslund J, Thomas M. The Emperors sham - wrong assumption that sham needling is sham. Acupunct Med. 2008 Dec;26(4):239-42. doi: 10.1136/aim.26.4.239. PMID 19098696
- [Background] Moffet HH. Sham acupuncture may be as efficacious as true acupuncture: a systematic review of clinical trials. J Altern Complement Med. 2009 Mar;15(3):213-6. doi: 10.1089/acm.2008.0356. PMID 19250001
- [Background] Hammerschlag R. Methodological and ethical issues in clinical trials of acupuncture. J Altern Complement Med. 1998 Summer;4(2):159-71. doi: 10.1089/acm.1998.4.159. PMID 9628206
- [Background] White AR, Filshie J, Cummings TM; International Acupuncture Research Forum. Clinical trials of acupuncture: consensus recommendations for optimal treatment, sham controls and blinding. Complement Ther Med. 2001 Dec;9(4):237-45. doi: 10.1054/ctim.2001.0489. PMID 12184353
- [Background] Park JE, Ryu YH, Liu Y, Jung HJ, Kim AR, Jung SY, Choi SM. A literature review of de qi in clinical studies. Acupunct Med. 2013 Jun;31(2):132-42. doi: 10.1136/acupmed-2012-010279. Epub 2013 Mar 13. PMID 23486017